CLINICAL TRIAL: NCT04818567
Title: Frequency and Causes of Failed Endoscopic Retrograde Cholangio-Pancreatography in AL-Rajhi Endoscopy Unit
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Soha Mohie El Din Mohamed, Resident doctor, Assiut University
Other Study IDs: ERCP failure
Record Dates: First submitted 2021-03-24; First posted 2021-03-26 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: ERCP, Failure, Complications, Cannulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The failure can be traced backed to operator causes, technical causes and patient causes.

the most common etiology is cannulation failure. ERCP complications includes post-ERCP pancreatitis, perforation, bleeding, cholangitis and cholecystitis.

ELIGIBILITY:
Inclusion Criteria:

* All cases underwent ERCP in our center from 1st of January, 2013 to 1st of January. 2021 with any causes of jaundice or any indication for which ERCP was done.

Exclusion Criteria:

* incomplete data or missing files were excluded from this study

Ages: 6 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All cases underwent ERCP in our center
Sampling Method: Probability Sample
Enrollment: 196 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-05-30 (Estimated)

PRIMARY OUTCOMES:
Frequency and causes of failed Endoscopic Retrograde Cholangio-Pancreatography in AL-Rajhi endoscopy unit | 2 years